CLINICAL TRIAL: NCT01820429
Title: Residual Platelet Activity Despite Aspirin Utilization in Patients With Non ST Elevation Acute Coronary Syndromes: Comparison Between the Acute and Chronic Phases
Brief Title: Residual Platelet Activity Despite Aspirin Utilization in Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: INCORPA
Record Dates: First submitted 2012-07-10; First posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Heart Disease; Non ST-elevation Acute Coronary Syndromes
Keywords: Platelet aggregation; Aspirin
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- First 48 hours: Patients in the first 48 hours of non ST-elevation acute coronary syndromes.
- 3 months after discharge: Patients with 3 months after hospital discharge for non ST-elevation acute coronary syndromes.

SUMMARY:
The purpose of this study is to compare the response to aspirin in the acute phase with the late phase of an acute coronary syndrome.

DETAILED DESCRIPTION:
The purpose of this study is to compare, in the same population, the response to aspirin in the initial phase (first 48 hours) with the late phase (after 3 months of discharge)of a non ST elevation acute coronary syndrome (angina or acute myocardial infarction).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of acute coronary syndrome without ST segment elevation, in the first 48 hours after the onset of the clinical symptoms
* Regular use of aspirin for at least seven days.

Exclusion Criteria:

* Previous use, in the last 7 days, of another antiplatelet agent than aspirin
* Use of antivitamin K in the last 3 weeks
* Hemoglobin < 10g/dL and / or hematocrit < 30% or > 50%, platelets count < 100.000/mm3 or > 500.000/mm3, creatinine clearance < 30 mL / minute
* Killip class III or IV
* Need for vasopressor or inotropic parenteral medication at inclusion in the study
* Percutaneous coronary intervention within 30 days or CABG in the last 90 days prior to study entry
* Current malignancy
* Hematologic diseases
* Refusal to sign the inform consent form
* Unable to attend the second visit (follow-up) for any reason except for death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 patients diagnosed with non ST acute coronary syndrome (unstable angina and myocardial infarction without ST elevation), with up to 48 hours of evolution from the onset of symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Compare platelet aggregation between the first 48 hours and 3 months after discharge. | 3 months

SECONDARY OUTCOMES:
Relation between platelet aggregability and the composite endpoint of death, myocardial infarction, unstable angina and need for revascularization or hospitalization at 3 months after discharge. | 3 months
Relation between the atherosclerotic burden by coronary angiography with the platelet aggregation in the first 48 hours. | 48 hours
Relation between C reactive protein and interleukin -6 with levels of platelet aggregation. | first 48 hours and 3 months
Relation between platelet aggregation and the presence or absence of selected polymorphisms. | first 48 hours and 3 months
Platelet aggregation in respect to age, gender, glucose at hospital arrival, glycated hemoglobin, statin, PPI, current smokers, ACE inhibitors, type of ACS presentation. | first 48 hours and 3 months
  Cut point for age 65 y, for glycemia 125 mg/dL, for glycated hemoglobin 6%

CONTACTS AND LOCATIONS:
Overall Officials: Jose C Nicolau, MD, PhD, Study Chair — Instituto do Coração (Heart Institute) - Clinical Hospitals, University of São Paulo Medical School
Locations (1):
- Instituto do Coração (Heart Institute) - Clinical Hospitals, University of São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.incor.usp.br